CLINICAL TRIAL: NCT01950923
Title: Sildenafil Prior to Robotic Partial Nephrectomy to Improve Postoperative Renal Function: A Randomized, Placebo-Controlled Pilot Study
Brief Title: Sildenafil Citrate Before Surgery in Improving Kidney Function in Patients With Kidney Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00021729-1; NCI-2013-00988 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA012197 (NIH)
Record Dates: First submitted 2013-09-24; First posted 2013-09-26 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Kidney Tumor
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (sildenafil citrate) (Experimental): Patients receive sildenafil citrate PO before the initiation of standard robotic partial nephrectomy.
  Interventions: Drug: sildenafil citrate; Procedure: therapeutic conventional surgery
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO before the initiation of standard robotic partial nephrectomy.
  Interventions: Other: placebo; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: sildenafil citrate — Given PO
  Other Names: Viagra
  Arms: Arm I (sildenafil citrate)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Procedure: therapeutic conventional surgery — Undergo standard robotic partial nephrectomy

SUMMARY:
This randomized pilot clinical trial studies sildenafil citrate before surgery in improving kidney function in patients with kidney cancer. Sildenafil citrate may help protect the kidney from the side effects of surgery and improve kidney function after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess accrual, retention, and participation rates for patients receiving sildenafil (sildenafil citrate) compared to placebo in patients undergoing robotic partial nephrectomy (RPN) for a suspected renal malignancy.

SECONDARY OBJECTIVES:

I. To evaluate individual alterations in glomerular filtration rate (GFR) at 24 hours, 48 hours and one month following RPN and compare these to the placebo group.

II. To evaluate individual alterations in proteinuria at 24 hours, 48 hours, one month and three months following RPN and compare these to the placebo group.

III. To measure between-group differences in estimated blood loss and hemoglobin concentration at 24 hours following RPN.

IV. To describe individual changes in blood pressure measurements as noted in the preoperative holding area, throughout the procedure and in the post-anesthesia care unit.

V. To describe between-group variations in vasopressor support or intravenous fluid requirements during the operative procedure.

VI. To compare overall complication rates (within 90 days postoperatively) between groups.

VII. To obtain a preliminary effect size of sildenafil on change in GFR at three months following RPN.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive sildenafil citrate orally (PO) before the initiation of standard robotic partial nephrectomy.

ARM II: Patients receive placebo PO before the initiation of standard robotic partial nephrectomy.

After completion of study treatment, patients are followed up at 1 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo robotic partial nephrectomy for suspected renal malignancy
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with a history of coronary artery disease (including history of myocardial infarction or cardiac stents) or a history of inducible ischemic changes on any prior cardiac stress testing
* History of adverse reactions to any phosphodiesterase (PDE) inhibitor (PDE type 5 inhibitor [PDE5i])
* Any patient currently taking a PDE5i will be asked to refrain from use for one week prior to their surgery; patients who have used a PDE5i within 72 hours of surgery will be excluded
* Pregnant women are excluded from this study
* Patients with only one kidney

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Accrual rate | Up to 6 months
  Reasons for declining enrollment to the study will be documented on the Declined Participation Form at the time patients are presented with the study.
Retention rate | Up to 3 months
  Retention will be assessed by whether or not the patient attends his or her 1 and 3 month postoperative visits.
Participation rate | Up to 6 months
  Reasons for declining enrollment to the study will be documented on the Declined Participation Form at the time patients are presented with the study.

SECONDARY OUTCOMES:
Change in GFR | Baseline to up to 1 month
  Regression analysis will be used; the change will be modeled, with adjustment for baseline GFR, to assess difference in the two study groups.
Change in proteinuria | Baseline to up to 3 months
  Compared between the two study groups.
Estimated blood loss | At 24 hours after RPN
  Compared between the two study groups.
Hemoglobin concentration | At 24 hours after RPN
  Compared between the two study groups.
Changes in blood pressure measurements | Baseline to up to 2 days after RPN
  Compared between the two study groups.
Vasopressor support requirements during the operative procedure | During RPN
  Compared between the two study groups.
Intravenous fluid requirements during the operative procedure | During RPN
  Compared between the two study groups.
Overall complication rates | Up to 90 days after RPN
  Compared between the two study groups.
Preliminary effect size of sildenafil citrate on change in GFR | At 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Hemal, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States